CLINICAL TRIAL: NCT05170542
Title: A Single-arm, Phase II Study of Camrelizumab Combined With S-1 Maintenance After First-Line Induction Chemotherapy in Patients With HER2 Negative Advanced Gastric Cancer
Brief Title: The Neoadjuvant Treatment of Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, WangXiang, chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-Ⅱ-09
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Efficacy and Safty of Camrelizumab Plus S-1 Maintenance After First-line Induction Chemotherapy for GC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+S-1 (Experimental)
  Interventions: Drug: Camrelizumab+S-1

INTERVENTIONS:
Drug: Camrelizumab+S-1 — Camrelizumab: intravenous drip, fixed dose 200 mg, D1, repeated once every 3 weeks.

SUMMARY:
In this study, We investigated the efficacy and safty of camrelizumab combined with S-1 maintenance after first-line induction chemotherapy for GC. Patients without progressive disease after 4-6 weeks of first-line chemotherapy with SOX will be treated with camrelizumab combined with S-1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged from 18 to 75 years old;
2. Subjects with histologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastro-esophageal junction (GEJ);
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry;
4. Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
5. Estimated life expectancy of more than 3 months;
6. Adequate haematological, hepatic and renal functions defined by the protocol;
7. Negative blood pregnancy test at Screening for women of childbearing potential; Highly effective contraception for both male and female subjects if the risk of conception exists;

Exclusion Criteria:

1. Concurrent anticancer treatment such as chemotherapy, radiotherapy, targeted or immunotherapy;
2. Tumor shown to be human epidermal growth factor 2 plus (HER2+);
3. Previous malignant disease (other than gastric cancer) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, colorectal, breast);
4. Severe infection (e.g. need for intravenous antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or fever (>38.5%) of unknown reason occurred during the screening period/before the first administration；
5. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy)); The subjects with childhood asthma who had been completely relieved and did not need any intervention or vitiligo in adulthood could be included, but the subjects who needed bronchodilator for medical intervention could not be included;
6. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method), or co infection of hepatitis B and hepatitis C;
7. Used immunosuppressive drugs within 14 days before the first dose of study drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids;
8. Accination with live or live/attenuated viruses within 28 days of the first dose of camrelizumab and while on trial is prohibited except for administration of inactivated vaccines;
9. History of uncontrolled intercurrent illness including hypertension, active infection, diabetes or cardiac diseases or symptoms;
10. Prior organ transplantation, including allogeneic stem-cell transplantation； Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-24 (Estimated); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of randomization to a minimum of 42 months
  PFS is defined as time (in months) from date of randomization to the date of the first documentation of objective progressive disease (PD) or death due to any cause in the absence of documented PD (whichever occurs first). PFS will be determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on investigator response assessment.

SECONDARY OUTCOMES:
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | From the the first dose of study drug administration up to 28 days after the last dose of study drug administration, assessed up to 3.5 years
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 28 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.
Objective Response Rate（ORR） | From the start of randomization to a minimum of 42 months
  Assess ORR, defined as Investigator-assessed CR + PR, per RECIST 1.1.
Disease Control Rate (DCR) | Time Frame: From the start of randomization to a minimum of 42 months
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated.
Overall Survival（OS） | From the start of randomization to a minimum of 42 months
  OS is defined as the time (in months) from randomization to the date of death, regardless of the actual cause of the subject's death.

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Zhao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided